CLINICAL TRIAL: NCT02271334
Title: Evaluation of Pharmacokinetics and Safety of A006 in Healthy Volunteers (A Randomized, Double- or Evaluator-blinded, Single-dose, Four-arm, Crossover Pharmacokinetics (PK) Study in Healthy Adults)
Brief Title: Evaluation of Pharmacokinetics and Safety of A006 in Healthy Volunteers
Acronym: A006-D
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: API-A006-CL-D
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Asthma
Keywords: Asthma; Albuterol
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment T1 (Experimental): One inhalation of 110 mcg A006 DPI. Total 110 mcg
  Interventions: Drug: A006 DPI
- Treatment T2 (Experimental): One inhalation of 220 mcg A006 DPI. Total 220 mcg.
  Interventions: Drug: A006 DPI
- Treatment R1 (Active Comparator): One inhalation of 90 mcg Proventil® MDI. Total 90 mcg.
  Interventions: Drug: Proventil® MDI
- Treatment R2 (Active Comparator): Two inhalations of 90 mcg Proventil® MDI. Total 180 mcg
  Interventions: Drug: Proventil® MDI

INTERVENTIONS:
Drug: A006 DPI — Single dose 110 mcg, 1 inhalation
  Other Names: Albuterol; Albuterol DPI
  Arms: Treatment T1
Drug: A006 DPI — Single dose 220 mcg, 1 inhalation
  Other Names: Albuterol; Albuterol DPI
  Arms: Treatment T2
Drug: Proventil® MDI — Single dose 90 mcg, 1 inhalation
  Other Names: Proventil®
  Arms: Treatment R1
Drug: Proventil® MDI — Single dose 90 mcg, 2 inhalations
  Other Names: Proventil®
  Arms: Treatment R2

SUMMARY:
The objective of this study is to evaluate the pharmacokinetics (PK) and safety profiles of A006, an Albuterol dry powder inhaler (DPI), following a single dose of 110 mcg (T1) or 220 mcg (T2), in healthy male and female adult volunteers.

DETAILED DESCRIPTION:
This study is a randomized, double or evaluator-blinded, single dose, four-arm, crossover PK study in eighteen (18) healthy volunteers, both male and female adults, at 18-40 years of age.

All candidates will be screened and only those who satisfy all enrollment criteria will be enrolled into this study. Each study subject will participate in a screening visit and four (4) study visits with one (1) randomized study treatment given in each visit.

PK samples will be analyzed with an established LC/MS/MS method. An End-of-Study (EOS) safety evaluation will be conducted at the end of Study Visit-4.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy, male and female adults, 18-40 years of age at Screening;
* Having no clinically significant respiratory, cardiovascular and other systemic or organic illnesses;
* Body weight ≥ 50 kg for men and ≥ 45 kg for women, and BMI within the range of 18.5 - 30.0 kg/m2 inclusive;
* Sitting blood pressure ≤ 135/90 mmHg;
* Demonstrating negative HIV, HBsAg and HCV tests, alcohol and nine panel urine drug screen tests;
* Demonstrating proficiency in the use of DPI and MDI or able to be trained in the proper use of these devices;
* Demonstrating Peak Inspiratory Flow Rate (PIF) within 80-150 L/min (after training), for at least 2 times consecutively, with a maximum of 5 attempts;
* Having no known hypersensitivity to any ingredients of A006 and Proventil® MDI (Albuterol, sulfate, lactose, milk protein, HFA-134a, oleic acid, or ethanol). (Subjects must be able to tolerate at least one teaspoon of milk);
* Women of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control; and
* Having properly consented and satisfied all other inclusion/exclusion criteria as required for this protocol.

Exclusion Criteria:

* A smoking history of ≥ 5 pack-years, or having smoked within 6 months prior to Screening;
* Upper respiratory tract infections within 2 weeks, or lower respiratory tract infection within 4 weeks, prior to Screening;
* Previous history of asthma or COPD;
* Any current or recent respiratory conditions that, per investigator discretion, might significantly affect pharmacodynamic response to the study drugs, including cystic fibrosis, bronchiectasis, tuberculosis, emphysema, and other significant respiratory diseases;
* Concurrent clinically significant cardiovascular, hematological, renal, neurologic, hepatic, endocrine, psychiatric, malignant, or other illnesses that in the opinion of the investigator could impact on the conduct, safety and evaluation of the study;
* ECG at Screening and Visit-1 baseline expressed any single or multiple premature ventricular contractions (PVC);
* ECG at Screening and Visit-1 baseline with a QTc reading greater than 450ms;
* Use of prohibited drugs or failure to observe the drug washout restrictions; and
* Having been on other clinical drug/device studies or donated blood in the last 30 days prior to Screening.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2014-10 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Area Under the Curve of Drug Concentration versus Time (AUC[0-t]) | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  Subject PK blood samples will be taken prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period. PK samples will be analyzed using a validated test method. Area under the curve of the drug concentration versus time curve (AUC[0-t]) for each treatment period will be calculated using the trapezoidal rule.
Peak Plasma Concentration (C[max]) | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  Subject PK blood samples will be taken prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period. PK samples will be analyzed using a validated test method. Peak plasma concentration (C[max]) will be the highest concentration of Albuterol during each treatment period.
Time to Reach Peak Plasma Concentration (t[max]) | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  Subject PK blood samples will be taken prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period. PK samples will be analyzed using a validated test method. Time to reach peak plasma concentration (t[max]) will be the time it takes to reach the highest concentration of Albuterol during each treatment period.
Plasma Albuterol Concentrations at All Time Points | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  Subject PK blood samples will be taken prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period. PK samples will be analyzed using a validated test method. Plasma Albuterol concentrations at these time points will be reported during each treatment period.

OTHER OUTCOMES:
Systolic Blood Pressure (SBP) at Screening | Within 14 days prior to Day 1 (Visit 1)
  Subjects will have their vital signs, i.e., blood pressure and heart rate, measured during the Screening Visit to ensure they are generally healthy.
Systolic Blood Pressure (SBP) | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  Subject will have their vital signs, i.e., blood pressure and heart rate, measured prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period.
Diastolic Blood Pressure (DBP) at Screening | Within 14 days prior to Day 1 (Visit 1)
  Subjects will have their vital signs, i.e., blood pressure and heart rate, measured during the Screening Visit to ensure they are generally healthy.
Diastolic Blood Pressure (DBP) | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  Subject will have their vital signs, i.e., blood pressure and heart rate, measured prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period.
Heart Rate (HR) at Screening | Within 14 days prior to Day 1 (Visit 1)
  Subjects will have their vital signs, i.e., blood pressure and heart rate, measured during the Screening Visit to ensure they are generally healthy.
Heart Rate (HR) | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  Subject will have their vital signs, i.e., blood pressure and heart rate, measured prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period.
12-Lead ECG QT Intervals at Screening | Within 14 days prior to Day 1 (Visit 1)
  12-Lead ECGs will be performed to measure QT and QTc intervals during the Screening Visit to ensure absence of overt cardiac illnesses.
12-Lead ECG QT Intervals | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  12-Lead ECGs will be performed to measure QT and QTc intervals prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period.
12-Lead ECG QTc Intervals at Screening | Within 14 days prior to Day 1 (Visit 1)
  12-Lead ECGs will be performed to measure QT and QTc intervals during the Screening Visit to ensure absence of overt cardiac illnesses.
12-Lead ECG QTc Intervals | Within 30 minutes prior to dosing (baseline) to 8 hours post-dose
  12-Lead ECGs will be performed to measure QT and QTc intervals prior to dosing and at multiple time points, up to 8 hours after dosing during each treatment period.
Complete Blood Count (CBC) at Screening | Within 14 days prior to Day 1 (Visit 1)
  A CBC will be performed as part of the subject safety evaluations at screening.
Complete Blood Count (CBC) at End-of-Study | 4 hours post-dose at Visit 4 (within 6 weeks after Day 1 (Visit 1))
  A CBC will be performed as part of the End-of-Study subject safety evaluations at end-of-study.
Comprehensive Metabolic Panel (CMP) at Screening | Within 14 days prior to Day 1 (Visit 1)
  A CMP will be performed as part of the subject safety evaluations at screening.
Comprehensive Metabolic Panel (CMP) at End-of-Study | 4 hours post-dose at Visit 4 (within 6 weeks after Day 1 (Visit 1))
  A CMP will be performed as part of the End-of-Study subject safety evaluations at end-of-study.
Urinalysis at Screening | Within 14 days prior to Day 1 (Visit 1)
  Routine and microscopic urinalysis will be performed as part of the subject safety evaluations at screening.
Urinalysis at End-of-Study | 4 hours post-dose at Visit 4 (within 6 weeks after Day 1 (Visit 1))
  Routine and microscopic urinalysis will be performed as part of the End-of-Study subject safety evaluations at end-of-study.
Incidents of Pregnancy at Screening | Within 14 days prior to Day 1 (Visit 1)
  A urinary pregnancy test will be performed for women of child-bearing potential as a part of the Screening Visit evaluations to determine the eligibility of the subject for the study.
Incidents of Pregnancy at End-of-Study | 4 hours post-dose at Visit 4 (within 6 weeks after Day 1 (Visit 1))
  A urinary pregnancy test will be performed for women of child-bearing potential as a part of the End-of-Study safety evaluations to determine if a pregnancy had occurred during the study.
Serious Adverse Events | Signing of Informed Consent at Screening Visit to End-of-Study Visit, an expected average of 7 Weeks
  Adverse drug events (ADEs), whether observed by investigators or reported by the subjects, will be documented, evaluated, followed up, and treated if deemed necessary. According to FDA guidelines, a serious ADE will refer to any adverse drug experience occurring at any dose that results in any of the following outcomes: 1) death; 2) a life-threatening adverse drug experience; 3) inpatient hospitalization or prolongation of existing hospitalization; 4) persistent or significant disability/incapacity; 5) congenital anomaly/birth defect; 6) other important medical events that may jeopardize the subject or may require medical or surgical intervention to prevent one of the outcomes listed in this definition. ADEs will be followed until stabilized/resolved or 30 days from the date the subject has finished the study, whichever is sooner.
Other Adverse Events | Signing of Informed Consent at Screening Visit to End-of-Study Visit, an expected average of 7 Weeks
  Adverse drug events (ADEs), whether observed by investigators or reported by the subjects, will be documented, evaluated, followed up, and treated if deemed necessary. ADEs will be followed until stabilized/resolved or 30 days from the date the subject has finished the study, whichever is sooner.

CONTACTS AND LOCATIONS:
Overall Officials: Safety Monitor, Study Director — Amphastar Pharmeceuticals, Inc.
Locations (1):
- Amphastar Site 0035, Cypress, California, United States

REFERENCES:
- [Background] Lipworth BJ, Clark DJ. Lung delivery of salbutamol given by breath activated pressurized aerosol and dry powder inhaler devices. Pulm Pharmacol Ther. 1997 Aug;10(4):211-4. doi: 10.1006/pupt.1997.0093. PMID 9695144
- [Background] Ahrens RC. The role of the MDI and DPI in pediatric patients: "Children are not just miniature adults". Respir Care. 2005 Oct;50(10):1323-8; discussion 1328-30. PMID 16185368
- [Background] Goldstein DA, Tan YK, Soldin SJ. Pharmacokinetics and absolute bioavailability of salbutamol in healthy adult volunteers. Eur J Clin Pharmacol. 1987;32(6):631-4. doi: 10.1007/BF02456001. PMID 3653233
- [Background] Hindle M, Newton DA, Chrystyn H. Dry powder inhalers are bioequivalent to metered-dose inhalers. A study using a new urinary albuterol (salbutamol) assay technique. Chest. 1995 Mar;107(3):629-33. doi: 10.1378/chest.107.3.629. PMID 7874928